CLINICAL TRIAL: NCT03646994
Title: A Real World Study to Evaluate the Efficacy and Safety of First Line Crizotinib in ROS1-rearranged Non-squamous Non-small Cell Lung Cancer
Brief Title: Real World Study on First Line Crizotinib in ROS1 Rearranged Advanced Non-squamous Non-small Cell Lung Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hunan Province Tumor Hospital (Other)
Responsible Party: Principal Investigator, Yongchang Zhang, Professor, Hunan Province Tumor Hospital
Other Study IDs: CORE
Record Dates: First submitted 2018-08-23; First posted 2018-08-24 (Actual); Last update posted 2023-12-27 (Actual); Status verified 2023-12

CONDITIONS: Non-small Cell Lung Cancer
Keywords: Non-small Cell Lung Cancer; Crizotinib; ROS1 Rearranged
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Crizotinib

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — tissue sample and plasma DNA
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cohorts 1: ROS1 fusion positive NSCLC patients who received crizotinib
  Interventions: Drug: Crizotinib

INTERVENTIONS:
Drug: Crizotinib — Crizotinib Cap 250 mg po bid

SUMMARY:
This study was designed to explore the efficacy and safety of Crizotinib as a first-line treatment for advanced NSCLC with ROS1 rearrangement positive mutation in the real world, explore the new drug resistance mechanism of ROS1 under Crizotinib treatment and the consistency of plasma and tissue detection driving genes, and finally evaluate the mutation spectrum of plasma dynamic detection driving genes. In predicting the risk of disease progression.

DETAILED DESCRIPTION:
This is a research project involving patients in Medical Oncology Department of Affiliated Cancer Hospital of Xiangya School of Medicine Central South University. Retrospective study of 40 patients with advanced non-squamous non-small cell lung cancer (NSCLC) using Crizotinib ROS1 rearrangement positive mutation was conducted to observe the efficacy and safety of Crizotinib regimen in the real world.Exploratory research contents are as follows: 1. Consistency between tissue gene test (NGS) and plasma gene test (NGS) at the initial diagnosis; 2. Consistency between NGS and plasma gene test (NGS) at the progression of clozotinib treatment; 3. Drug resistance mechanism of clozotinib in ROS1 rearrangement positive NSCLC; 4. Plasma drug resistance. Large panel dynamic driven gene mutation analysis was used to construct disease progression risk model.

ELIGIBILITY:
Inclusion Criteria:

* ≥18，Advanced Non-squamous Non-small Cell Lung Cancer Confirmed by Histopathology
* ROS1 Arranged Positive
* ROS1 Arranged Detection Method is NGS
* First Diagnosis and Treatment
* Treatment Plan is Kazolinib 250mg po bid

Exclusion Criteria:

* Patients received antitumor treatment before
* Patients with contraindication of chemotherapy
* Pregnant or breast feeding women

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: ROS1 rearranged Advanced Non-squamous Non-small Cell Lung Cancer Confirmed by NGS
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2018-08-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
PFS | may 2018- may 2019 (1 year)
  progression survival time

SECONDARY OUTCOMES:
ORR | may 2018- may 2019 (1 year)
  objective response rate
OS | may 2018- may 2019 (1 year)
  over survival time

CONTACTS AND LOCATIONS:
Overall Officials: Yongchang Zhang, MD, Principal Investigator — Hunan Cancer Hospital
Locations (1):
- Hunan Cancer Hospital, Changsha, Hunan, China

REFERENCES:
- [Derived] Zhang Y, Zhang X, Zhang R, Xu Q, Yang H, Lizaso A, Xu C, Liu J, Wang W, Ou SI, Zhang J, Song Z, Yang N. Clinical and molecular factors that impact the efficacy of first-line crizotinib in ROS1-rearranged non-small-cell lung cancer: a large multicenter retrospective study. BMC Med. 2021 Sep 13;19(1):206. doi: 10.1186/s12916-021-02082-6. PMID 34511132